CLINICAL TRIAL: NCT01614509
Title: Combined Therapy of Posterior Subtenon Triamcinolone Acetonide and Intravitreal Bevacizumab for Macular Edema Secondary to Branch Retinal Vein Occlusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeungnam University College of Medicine (Other)
Responsible Party: Principal Investigator, Min Sagong, Assistant Professor, Yeungnam University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCR-11-144
Record Dates: First submitted 2012-06-05; First posted 2012-06-08 (Estimated); Results first posted 2012-12-04 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Branch Retinal Vein Occlusion
Keywords: branch retinal vein occlusion; bevacizumab; triamcinolone acetonide
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monotherapy group (Experimental): The monotherapy group receive intravitreal injection of 1.25 mg/0.05 ml bevacizumab. The injections are performed using 0.5% proparacaine drops for topical anesthesia under sterile conditions. The bevacizumab is injected through the pars plana using a 30-gauge needle.
  Interventions: Procedure: intravitreal bevacizumab monotherapy
- Combined group (Experimental): The combined group receive intravitreal injection of 1.25 mg/0.05 ml bevacizumab and posterior subtenon injection of 40 mg/1.0 ml triamcinolone acetonide. The injections are performed using 0.5% proparacaine drops for topical anesthesia under sterile conditions. The Bevacizumab is injected through the pars plana using a 30-gauge needle and triamcinolone acetonide is injected through the posterior subtenon area (near macula) by using a 27-gauge needle at the same time.
  Interventions: Procedure: combined therapy of posterior subtenon triamcinolone acetonide and intravitreal bevacizumab injection

INTERVENTIONS:
Procedure: intravitreal bevacizumab monotherapy — The monotherapy group receive intravitreal injection of 1.25 mg/0.05 ml bevacizumab. The injections are performed using 0.5% proparacaine drops for topical anesthesia under sterile conditions. The bevacizumab is injected through the pars plana using a 30-gauge needle.
  Arms: Monotherapy group
Procedure: combined therapy of posterior subtenon triamcinolone acetonide and intravitreal bevacizumab injection — The combined group receive intravitreal injection of 1.25 mg/0.05 ml bevacizumab and posterior subtenon injection of 40 mg/1.0 ml triamcinolone acetonide. The injections are performed using 0.5% proparacaine drops for topical anesthesia under sterile conditions. The bevacizumab is injected through the pars plana using a 30-gauge needle and triamcinolone acetonide is injected through the posterior subtenon area (near macula) by using a 27-gauge needle at the same time.
  Arms: Combined group

SUMMARY:
This study compares the efficacy of intravitreal bevacizumab monotherapy only or combined therapy of posterior subtenon's triamcinolone acetonide and intravitreal bevacizumab for the treatment of macular edema associated with branch retinal vein occlusion.

ELIGIBILITY:
Inclusion Criteria:

1. The participant must have macular edema associated branch retinal vein occlusion.
2. The participant has retinal photographs, optical coherence tomography (OCT) and angiography of sufficient quality, allowing assessment of the macular area according to standard clinical practice.
3. The participant must be willing and able to comply with the protocol.

Exclusion Criteria:

1. The participant has BRVO with other ocular vascular diseases such as central retinal vein occlusion, hypertensive retinopathy, etc.
2. The participant has any additional ocular diseases that have irreversibly compromised or could likely compromise the visual acuity of the study eye including amblyopia, anterior ischemic optic neuropathy, clinically significant diabetic macular edema, severe non proliferative diabetic retinopathy, or proliferative diabetic retinopathy.
3. The participant has a history of treatment for BRVO in the study eye with focal laser photocoagulation, intravitreal triamcinolone acetonide injection or intravitreal Bevacizumab injection
4. The participant has a history of intraocular surgery (including lens replacement surgery).
5. The participant has a history of ocular trauma, or current ocular or periocular infection (including any history of ocular herpes zoster or simplex).

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Yeungnam University College of Medicine, Daegu, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Conditions: Macular edema secondary to Branch Retinal Vein Occlusion The recruitment period: from Jan 2012 to Aug 2012
Pre-assignment Details: During the follow up period, Not attendants, participants who were received other intraocular surgeries and etc. were excluded.
Period: Overall Study
Arm/Group | Monotherapy Group | Combined Group
Started | 24 | 21
Completed | 23 | 18
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Monotherapy Group | Combined Group | Total
Number analyzed (Participants) | 24 | 21 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 10 | 7 | 17
Age Continuous [Mean (Standard Deviation); unit: years] | 62.04 (10.498) | 60.24 (14.983) | 61.20 (12.668)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 14 | 11 | 25
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 24 | 21 | 45

OUTCOME MEASURES:

1. Secondary Outcome: Additional Intravitreal Bevacizumab Injection
Description: Comparison of the additional intravitreal bevacizumab injection of intravitreal bevacizumab monotherapy or combined therapy of posterior subtenon triamcinolone acetonide and intravitreal bevacizumab during 6 months
Time Frame: 6 months
Population: We evaluated mean times of additional intravitreal injection because of recurrent macular edema within participants who who were finished 6 months follow up periods.
Measure: Mean (Standard Deviation); unit: times of injection
Arm/Group | Monotherapy Group | Combined Group
Number analyzed (Participants) | 23 | 18
times of injection | 0.96 (0.83) | 0.44 (0.70)

2. Primary Outcome: Changes of Central Retinal Thickness
Description: Changes of central retinal thickness on optical coherence tomography (OCT) at baseline and 1, 3, 6 month after injection
Time Frame: baseline, 1, 3, 6 months after injection
Population: Participants who were finished 6 months follow up period.
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | Monotherapy Group | Combined Group
Number analyzed (Participants) | 23 | 18
micrometer
  at baseline | 510.35 (185.36) | 468.22 (159.26)
  1 month after injection | 291.48 (100.19) | 233.33 (79.95)
  3 months after injection | 265.35 (106.85) | 233.22 (57.09)
  6 months after injection | 246.48 (88.00) | 217.83 (42.64)
Statistical Analysis 1: Comparison: Monotherapy Group vs Combined Group; Central retinal thickness was measured using an optical coherence tomography by every visit. And we compare the difference of central retinal thickness between two groups; Test type: Non-Inferiority or Equivalence — Central retinal thickness was measured using an optical coherence tomography by every visit intended for all participants; p = 0.60, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Monotherapy Group | Combined Group
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/21
Other Adverse Events (participants affected / at risk) | 0/24 | 0/21

LIMITATIONS AND CAVEATS:
The limitation of our study include short duration of follow up (6 months) and small populations of study enroll (45 patients)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No